CLINICAL TRIAL: NCT03503370
Title: Preventing Diabetic Foot Ulcers Through Manipulating the Skin Microbiota
Brief Title: Preventing Diabetic Foot Ulcers Through Cleaner Feet
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: INFB-015-17F
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Foot Ulcer
Keywords: topical chlorhexidine; prevention; clinical trial
MeSH Terms: conditions — Diabetic Foot | interventions — Chlorhexidine

STUDY DESIGN:
Intervention Model Description: This is a single center, randomized, double blind (participant, outcome assessor), parallel group clinical trial comparing daily foot care with cloths containing 2% chlorhexidine compared to daily foot care with cloths not containing chlorhexidine.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chlorhexidine (Experimental): Participants randomized to the intervention will wash their feet using 2% CHLORHEXIDINE GLUCONATE CLOTHS to wipe down their feet each day and then apply supplied chlorhexidine-compatible over-the-counter moisturizer.
  Interventions: Drug: Chlorhexidine
- Placebo (Placebo Comparator): Participants randomized to the placebo will wash their feet using COMFORT BATH CLOTHS to wipe down their feet each day and then apply supplied chlorhexidine-compatible over-the-counter moisturizer.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chlorhexidine — Participants randomized to the intervention will wash their feet using 2% CHLORHEXIDINE GLUCONATE CLOTHS to wipe down their feet each day and then apply supplied chlorhexidine-compatible over-the-counter moisturizer.
  Arms: Chlorhexidine
Drug: Placebo — Participants randomized to the placebo will wash their feet using COMFORT BATH CLOTHS to wipe down their feet each day and then apply supplied chlorhexidine-compatible over-the-counter moisturizer.
  Arms: Placebo

SUMMARY:
Foot complications are among the most serious and costly complications of diabetes. People with diabetes have a 10-fold increased risk for a leg or foot amputation compared to those that do not have diabetes. Amputation of all or part of foot is usually preceded by a foot ulcer, which became infected. This is a clinical trial to test the effectiveness of a topical antiseptic, chlorhexidine, for daily foot cleaning on the occurrence of diabetic foot ulcers in Veterans at high risk of a diabetic foot ulcer.

DETAILED DESCRIPTION:
Population: Up to 200 Veterans at high risk of a diabetic foot ulcer

Site: VA Maryland Health Care System (VAMHCS)

Study Duration: Approximately 5 years

Study Design: Randomized double-blind clinical trial comparing a) a daily foot care regimen with cloths containing 2% chlorhexidine to b) a daily foot care regimen with cloths not containing 2% chlorhexidine

Objectives:

Primary: To determine if chlorhexidine reduces the occurrence of foot complications including chronic foot ulcer, foot infection or foot amputation.

Secondary: To determine if chlorhexidine increases antibiotic resistance among bacterial pathogens on feet.

Exploratory: To describe changes in the microbiota of the feet with chlorhexidine and foot complications

Treatment Regimens: 2% Chlorhexidine Gluconate Cloths versus Bath Cloths

Route of Administration: Topical application on the feet

Dose and Interval: 1 cloth daily

Duration of Participant's Participation: Up to 13 months

ELIGIBILITY:
Inclusion Criteria:

* Adults >=18 years
* Clinical diagnosis of diabetes
* At high risk for a new diabetic foot ulcer due to: 1)Past history of diabetic foot ulcer or 2)Past history of major foot surgery including partial foot amputation or 3)Past history of major foot infection or 4)Neuropathy and onychomycosis and hemoglobin A1C >8% or 5)Neuropathy and peripheral vascular disease or 6)Dialysis or 7)Past history of Charcot foot or 8)Past history of peripheral vascular surgery or angiography with stent
* Two feet (can have amputation of part of the foot)
* At least one foot without a foot ulcer
* Permanent mailing address suitable for provision of specimen collection materials and telephone suitable for monthly follow-up
* Able to give written informed consent

Exclusion Criteria:

* Amputation of the foot planned to treat current foot ulcer or wound
* Current foot infection
* Use of topical chlorhexidine on feet 7 days prior to randomization
* History of an allergic reaction to chlorhexidine
* Unable to use wipes for foot care
* Inability to walk
* Life expectancy less than 12 months
* Plans to move out of the area in the next 13 months
* Requires equivalent of institutional care (e.g. nursing home)
* Any other criteria which, in the investigator's opinion, would compromise the safety of the study, the ability of a subject to participate, or the results of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Claire Roghmann, MD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Final data sets underlying all publications resulting from the proposed research will be shared outside VA. A limited dataset will be created and shared pursuant to a Data Use Agreement. Final data sets will be maintained locally until enterprise-level resources become available. Upon request, we will provide an electronic limited dataset to others in the scientific community with the implementation of appropriate data use agreements.
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol and statistical analysis plan are available now on the CT.gov page for this study. Final datasets underlying all publications will be made available upon publication of each paper.
Access Criteria: Implementation of appropriate data use agreements. Email the study PI, Dr. Mary-Claire Roghmann (mroghmann@som.umaryland.edu), to start the process.

REFERENCES:
- [Derived] Lydecker AD, Kim JJ, Robinson GL, Johnson JK, Brown CH, Petruccelli CC, Terrin ML, Margolis DJ, Roghmann MC. Chlorhexidine vs Routine Foot Washing to Prevent Diabetic Foot Ulcers: A Randomized Clinical Trial. JAMA Netw Open. 2025 Feb 3;8(2):e2460087. doi: 10.1001/jamanetworkopen.2024.60087. PMID 39964684

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between January 2019 and December 2021 in the Baltimore VA Medical Center.
Period: Overall Study
Arm/Group | Chlorhexidine | Placebo
Started | 88 | 87
Completed | 85 | 86
Not Completed | 3 | 1
Not completed — Death | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chlorhexidine | Placebo | Total
Number analyzed (Participants) | 88 | 87 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (8) | 68 (10) | 68 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 85 | 85 | 170
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 87 | 87 | 174
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 60 | 57 | 117
  White | 25 | 28 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 88 | 87 | 175
Healed foot complication [Count of Participants; unit: Participants] — Healed foot complication is defined as a chronic foot ulcer, a major foot infection or a partial foot amputation that has healed prior to the study randomization visit. The healed foot complication could be on either foot.
  Participants | 48 | 43 | 91

OUTCOME MEASURES:

1. Primary Outcome: Time to New Foot Complication Among All Randomized Participants
Description: Time in days to new foot complication (analyzed with the use of unadjusted Cox proportional-hazard models to identify time to new foot complication; the results we are reporting are number of participants who developed a new foot complication in the 12 months post randomization). A new foot complication is defined as either 1) a new chronic (present 28 days from initial diagnosis) foot ulcer or wound or 2) a moderate or severe foot infection (as defined by IDSA Diabetic Foot Infection Severity classification: Table 2) not from an existing ulcer or 3) a foot amputation for a new ulcer.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine | Placebo
Number analyzed (Participants) | 88 | 87
Participants | 12 | 14
Statistical Analysis 1: Comparison: Chlorhexidine vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.39 to 1.80] — Hazard ratio from Cox Proportional Hazard comparing the chlorhexidine group to the placebo group

2. Secondary Outcome: Susceptibility to Chlorhexidine Among Bacterial Pathogens on the Feet
Description: Susceptibility to chlorhexidine among bacterial pathogens on the feet. Chlorhexidine minimum inhibitory concentration (MIC) values were normalized across pathogens by subtracting the median MIC value (MIC50) from the literature for each pathogen from the observed MIC value on a log2() scale. The results we are reporting are the mean normalized MIC values and the Wilcoxon Rank Sum test comparing the difference in distribution of normalized MIC values. Effect size is expressed in means as this is more sensitive to group differences than the median. The possible range for the normalized observed MIC values on a log2() scale is from -8 to 8 with a higher value indicating that the pathogens collected were more resistant to chlorhexidine as compared to the median MIC values reported in the literature.
Time Frame: 4 weeks after stopping the intervention (approximately 13 months after randomization)
Population: Participants must have at least one bacterial pathogen on their feet to be included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chlorhexidine | Placebo
Number analyzed (Participants) | 27 | 28
units on a scale | -1.83 (1.44) | -1.88 (1.52)
Statistical Analysis 1: Comparison: Chlorhexidine vs Placebo; Test type: Superiority; p = 0.97, Wilcoxon (Mann-Whitney)

3. Other Pre Specified Outcome: Time to New Foot Complication Among Participants With a Healed Foot Complication at Randomization.
Description: as for outcome 1
Time Frame: 12 months
Population: Participants must have had a healed foot complication at randomization to be included.
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine | Placebo
Number analyzed (Participants) | 48 | 43
Participants | 11 | 12
Statistical Analysis 1: Comparison: Chlorhexidine vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.34 to 1.77] — Hazard ratio from Cox Proportional Hazard comparing the chlorhexidine group to the placebo group

ADVERSE EVENTS:
Time Frame: Adverse events were actively assessed from the enrollment visit until the final study visit for each participant. The time from enrollment visit to final study visit was typically 13 months for a given participant. Enrollment began in January 2019 and the final study visit occurred in December 2022.
Description: Participants were asked about adverse events on a monthly basis.
Arm/Group | Chlorhexidine | Placebo
All-Cause Mortality (participants affected / at risk) | 3/88 | 1/87
Serious Adverse Events (participants affected / at risk) | 23/88 | 17/87
Other Adverse Events (participants affected / at risk) | 1/88 | 2/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chlorhexidine (N=88) | Placebo (N=87)
Anemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Brain aneurysm (Nervous system disorders) | 1 | 0
COVID-19 (Infections and infestations) | 3 | 1
Cellulitis (Infections and infestations) | 2 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Cervical radiculopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest pain, NOS (Cardiac disorders) | 0 | 1
Concussion (Nervous system disorders) | 0 | 1
Congestive heart failure (Cardiac disorders) | 3 | 2
Dehydration (General disorders) | 0 | 1
Diabetic foot infection (Infections and infestations) | 4 | 5
External ear infection (Infections and infestations) | 1 | 0
Fall due to general weakness (General disorders) | 1 | 0
Gallstone pancreatitis (Gastrointestinal disorders) | 0 | 1
Gout (Musculoskeletal and connective tissue disorders) | 1 | 0
Hyperglycemia (Gastrointestinal disorders) | 1 | 0
Hyperkalemia (Renal and urinary disorders) | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 1
Kidney transplant (Renal and urinary disorders) | 1 | 0
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Muscle weakness, NOS (General disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Near syncope, NOS (General disorders) | 0 | 1
Near syncope, NOS (Nervous system disorders) | 1 | 1
Opioid Use Disorder (Psychiatric disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2
Transient Ischemic Attack (Nervous system disorders) | 1 | 0
(General disorders) | 1 | 0
Urinary track infection (Infections and infestations) | 2 | 1
Weakness, NOS (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chlorhexidine (N=88) | Placebo (N=87)
Diabetic foot infection (Infections and infestations) | 0 | 1
Fall due to knee weakness (General disorders) | 1 | 0
Vaccine side effects (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT03503370/Prot_001.pdf
  • Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT03503370/SAP_000.pdf